CLINICAL TRIAL: NCT04515134
Title: Follicular Fluid Coenzyme Q10 Level in Women Undergoing Intracytoplasmic Sperm Injection
Brief Title: Assessment of Follicular Fluid Level of Coenzyme Q10 in Women Undergoing ICSI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Mohamed Atef Mohamed, doctor, South Valley University
Other Study IDs: follicular fluid Coenzyme Q10
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Pregnancy Outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — follicular fluid of the ovary will be aspirated, centrifuged and assessed for coenzyme Q10
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: assessment of follicular level of coenzyme Q10 in the ovaries in females undergoing ICSI — human coenzyme Q10 (CoQ10) ELISA kit

SUMMARY:
The aim of this study to assess the follicular fluid level of coenzyme Q10 in women undergoing intracytoplasmic sperm injection (ICSI) and its impact on pregnancy outcome.

DETAILED DESCRIPTION:
ICSI was first applied to human gametes in 1988, it was first used in cases of fertilization failure after standard IVF or when few sperm cells were available. The first pregnancies were reported in Belgium in 1992.It is a part of an in vitro fertilization (IVF) cycle and refers to a technique in which a single sperm is injected directly into the cytoplasm of a mature oocyte (Palermo et al.,1992).

Oocyte quality remains the most important issue during in vitro fertilization (IVF) cycles, it is affected mainly by age of woman and ovarian reserve (Trifunovic et al., 2004).

Oocyte maturation is a complex process including nuclear and cytoplasmic components. Mitochondria which is in the cytoplasm is the key regulator of energy production via oxidative phosphorylation process which is extremely important in oocyte maturation process. Any problem during oxidative phosphorylation might affect both the quality and DNA content of the oocytes (Ben-Meir et al., 2015).

Oxidative phosphorylation involves the action of the mitochondrial respiratory chain which consists of four complexes that are located in the inner mitochondrial membrane (May-Panloup et al., 2007). These are the NAD-linked dehydrogenase, Flavoproteins, Co-enzyme Q10, and cytochromes. Coenzyme Q10 (Ubiquinone) is structurally similar to vitamin E and vitamin K. It acts as a carrier of proton (H+) from flavoproteins to cytochrome (Bentinger et al., 2007).

Coenzyme Q10 is essential for stability and action of complex III (May-Panloup et al., 2007). It also participates in the transport of protons in the mitochondria to maintain the membrane potential and drive ATP formation through ATP synthetase so it has a critical role in cell growth and energy metabolism. One of the most important factors during oogenesis and oocyte maturation is energy consumption so CoQ10 was reported to improve development, hatching, cell proliferation, and ATP content of in vitro-produced bovine embryos (Gendelman et al., 2012; Stojkovic et al., 1999).

Coenzyme Q10 is a commonly used antioxidant supplement in multiple clinical conditions like diabetes, cancer, and cardiovascular diseases. Also, it was shown that Coenzyme Q10 improves sperm motility, semen quality, and pregnancy rate (Garrido-Maraver et al., 2014). Recently Bentov et al. reported that the use of coenzyme Q10 supplementation resulted in reduced aneuploidy and increased pregnancy rate however it is not clinically significant (Bentov et al., 2014).

Several studies reported that pretreatment with CoQ10 could improve ovarian response to stimulation and embryological parameters in women with poor ovarian reserve in IVF-ICSI cycles, however their results are conflicting so further work is needed to determine whether there is an effect on clinical endpoints (Akarsu et al., 2017). In our study we will investigate the relationship between follicular fluid level of Coenzyme Q10 and clinical pregnancy rate (Xu et al., 2018).

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 20-42 years.
2. Normal and Poor responders women undergoing ICSI procedure.

Exclusion Criteria:

1. Hyper responder patients as polycystic ovarian syndrome (PCOs) patients.
2. Endocrine or metabolic diseases including hyperprolactinoma, hypothyroidism and hyperthyroidism, DM and adrenal disease
3. Patients with severe male factor or Y chromosome abnormality.
4. Patients with systemic disease such as chronic renal disease, chronic liver disease and systemic lupus disease.
5. patients with uterine cavity pathology or abnormality (endometrial polyp, myoma, hyperplasia, congenital abnormality) detected by trasvaginal 3-dimentional ultrasound or office hysteroscopy.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This work will be conducted on normal and poor responder women undergoing ICSI procedure in ART unit in Obstetrics and Gynaecology department, South Valley University hospital female patient aged 20-42 years.
  poor responders have at least 2 of the following features:
  1. advanced maternal age (40 years or more).
  2. previous poor ovarian response (3 or less oocyte retrieved following stimulation).
  3. abnormal ovarian reserve teseting (AFC 5-7 or AMH 0.5-1).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-08-05 (Estimated); Study Completion 2022-09-10 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | baseline
  clinical pregnancy rate following the intracytoplasmic sperm injection (ICSI) and its relation to follicular fluid coenzyme Q10.

SECONDARY OUTCOMES:
implantation rate | baseline
  Implantation rate and assessment of embroys quality according to Istanbul consensus for embryo quality assessment (Balban et al., 2011).

CONTACTS AND LOCATIONS:
Overall Officials: mahmoud s mowad, MD, Study Chair — South Valley University
Locations (1):
- Mohamed Mohamed Atef, Alexandria, aAlexandria, Egypt

REFERENCES:
- [Background] Akarsu S, Gode F, Isik AZ, Dikmen ZG, Tekindal MA. The association between coenzyme Q10 concentrations in follicular fluid with embryo morphokinetics and pregnancy rate in assisted reproductive techniques. J Assist Reprod Genet. 2017 May;34(5):599-605. doi: 10.1007/s10815-017-0882-x. Epub 2017 Feb 9. PMID 28185121
- [Background] Ben-Meir A, Burstein E, Borrego-Alvarez A, Chong J, Wong E, Yavorska T, Naranian T, Chi M, Wang Y, Bentov Y, Alexis J, Meriano J, Sung HK, Gasser DL, Moley KH, Hekimi S, Casper RF, Jurisicova A. Coenzyme Q10 restores oocyte mitochondrial function and fertility during reproductive aging. Aging Cell. 2015 Oct;14(5):887-95. doi: 10.1111/acel.12368. Epub 2015 Jun 26. PMID 26111777
- [Background] Bentov Y, Hannam T, Jurisicova A, Esfandiari N, Casper RF. Coenzyme Q10 Supplementation and Oocyte Aneuploidy in Women Undergoing IVF-ICSI Treatment. Clin Med Insights Reprod Health. 2014 Jun 8;8:31-6. doi: 10.4137/CMRH.S14681. eCollection 2014. PMID 24987272
- [Background] Alpha Scientists in Reproductive Medicine and ESHRE Special Interest Group of Embryology. The Istanbul consensus workshop on embryo assessment: proceedings of an expert meeting. Hum Reprod. 2011 Jun;26(6):1270-83. doi: 10.1093/humrep/der037. Epub 2011 Apr 18. PMID 21502182